CLINICAL TRIAL: NCT06489522
Title: Supporting the Implementation of a Parenting Intervention for Mothers With Substance Use Disorder in the Pediatric Medical Home
Brief Title: Parenting Intervention for Mothers With Substance Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-44513
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Substance Use Disorders; Children of Mothers With Substance Use Disorders
Keywords: Parent Child Interaction Therapy (PCIT); Effective parenting skills; THRIVE; SOFAR clinic; Boston Medical Center
MeSH Terms: conditions — Substance-Related Disorders | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: Approximately 10 high-risk mother-child dyads (defined as a mother having an episode of relapse in the past two years) and approximately 10 low-risk mother-child dyads (defined as mother not having any episodes of relapse in the past two-years) will be enrolled. There will be 1 therapist and 9 clinical stakeholders (Patient Navigators, program manager, pediatricians, peer recovery coaches involved in the care of mother-child dyads in the SOFAR Program).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Threat, harm, risk, investigation, vulnerability and engagement (THRIVE) intervention (Experimental): The THRIVE intervention will be offered by a trained therapist to participants (mother-child dyads) in the SOFAR Clinic.
  Interventions: Behavioral: THRIVE

INTERVENTIONS:
Behavioral: THRIVE — THRIVE is a brief, parent child interaction therapy (PCIT) based telehealth intervention delivered over 6-sessions that has been tested in pediatric and community-based settings.

SUMMARY:
Children of mothers with substance use disorder (SUD) constitute a growing and highly vulnerable population. Evidence-based parenting interventions have the potential to both support parents' recovery and mental health by helping them cope with stress of parenthood and promote the optimal development of their children by supporting responsive parenting. The Supporting Our Families through Addiction and Recovery (SOFAR) pediatric medical home for families and children impacted by SUDs, with integrated behavioral health (IBH), provides an opportune setting for addressing the needs of mothers and children impacted by SUDs. While many families are thriving in the program, there is a strong unmet need for evidence-based parent-training interventions, particularly during the preschool period.

This study aims to evaluate the implementation of a brief, parent child interaction therapy (PCIT)-based intervention, entitled Threat, harm, risk, investigation, vulnerability and engagement (THRIVE), that will be offered in the SOFAR Clinic at Boston Medical Center. THRIVE is a safe, 6-session telehealth intervention that has been tested in pediatric and community-based settings. The evidence-based suggests that THRIVE is associated with significant improvements in child behaviors and parenting stress.

The investigators hypothesize that offering THRIVE through the SOFAR pediatric primary care program will be feasible and acceptable, improving access to and engagement in evidence-based parenting interventions among mothers with substance use disorder who receive parenting support through our integrated behavioral health model. In addition to studying the implementation of this evidence-based intervention, this study will allow the researchers to test data collection procedures (pre and post-interventions assessments) to inform a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* English speaking
* ≥ 18 years of age
* Mother to an index child between 3 years, 0 months to 6 years, 11 months of age who receives primary care at Boston Medical Center
* Primary caregiver to the index child,
* Engaged in formal SUD recovery supports (e.g., medication for opioid use disorder, support groups specific to people in recovery and falls into one of these two enrollment groups: A) "high-risk" substance use disorder defined >=1 episode of relapse within the past two years OR B) "low-risk" defined as zero episodes of relapse within the past two years.

Children:

* Between 3 years, 0 months to 6 years, 11 months of age,
* Enrolled mother is primary caregiver.

THRIVE Therapist:

* Embedded social worker in the SOFAR program delivering the THRIVE intervention

Clinical Stakeholders:

* Patient Navigators, program manager, pediatricians, peer recovery coaches involved in the care of mother-child dyads in the SOFAR Program.

Exclusion Criteria:

Mothers:

* Has an index child who has complex medical problems (e.g., autism spectrum disorder) that significantly impact the child's ability to interact with the parent (determination by child's primary care pediatrician)
* Severe cognitive limitation or medical or psychiatric condition that limits their capacity to provide informed consent
* Concurrent participation in another parent training intervention

Children:

* Has any complex medical problems (as assessed by their pediatrician) that significantly impact the child's ability to interact with the mother.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the THRIVE intervention | 12 months
  The Therapy Attitude Inventory survey will be used to collect assess mother/birthing parent acceptability of the THRIVE intervention. It is a 16 item instrument with 5 potential response per Question. Scores can range from 16 to 80 and higher scores are associated with higher acceptability.
Fidelity of the THRIVE intervention | 12 months
  The Treatment Integrity Checklist will be used to assess fidelity. It will be completed by research staff via review of video-recorded THRIVE sessions to monitor adherence to THRIVE core components.
Feasibility of the THRIVE intervention based on enrollment | 12 months
  The number of families ineligible, approached, and enrolled will be documented from study records.
Total number of THRIVE intervention sessions | 12 months
  The total number of sessions completed will be abstracted from the study records.
Duration of THRIVE intervention sessions | 12 months
  The duration of the sessions will be documented in minutes.
Percent of days homework completed | 12 months
  Percent of days homework completed will be obtained from study records
Feasibility of the THRIVE intervention based on retention | 12 months
  Retention will be assessed by the time to loss of follow-up.
Perceived reasons for discontinuation of THRIVE | 12 months
  The perceived reasons for discontinuation will be documented in the study records.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Elansary, MD MPhil, Principal Investigator — Boston Medical Center, Pediatrics
Locations (1):
- Boston Medical Center, SOFAR Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No